CLINICAL TRIAL: NCT03731364
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 (Vocacapsaicin) in Subjects Undergoing Total Knee Arthroplasty
Brief Title: Study of CA-008 (Vocacapsaicin) in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concentric Analgesics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA-PS-203
Record Dates: First submitted 2018-10-24; First posted 2018-11-06 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-12

CONDITIONS: Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CA-008 5 mg (0.05 mg/mL) Cohort 1 (Active Comparator): Cohort 1 (5 mg), was prepared at 0.05 mg/mL CA-008 (vocacapsaicin)
  Interventions: Drug: CA-008
- Placebo - Cohort 1 (Placebo Comparator): Placebo for Cohort 1
  Placebo comparator identical in appearance to the investigational product, containing the same excipients as the active
  Interventions: Drug: Placebo
- CA-008 10 mg (0.1 mg/mL) Cohort 2 (Active Comparator): Cohort 2 (10 mg), was prepared at 0.1 mg/mL CA-008 (vocacapsaicin)
  Interventions: Drug: CA-008
- CA-008 15 mg (0.15 mg/mL) Cohort 3 (Active Comparator): Cohort 3 (15 mg), was prepared at 0.15 mg/mL CA-008 (vocacapsaicin)
  Interventions: Drug: CA-008
- Placebo - Cohorts 2 and 3 (Placebo Comparator): Placebo - Cohorts 2 and 3
  Placebo comparator identical in appearance to the investigational product, containing the same excipients as the active
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CA-008 — 5 mg CA-008 (0.05 mg/mL), 10 mg CA-008 (0.1 mg/mL) and 15 mg CA-008 (0.15 mg/mL)
  Other Names: vocacapsaicin
  Arms: CA-008 10 mg (0.1 mg/mL) Cohort 2; CA-008 15 mg (0.15 mg/mL) Cohort 3; CA-008 5 mg (0.05 mg/mL) Cohort 1
Drug: Placebo — Placebo
  Arms: Placebo - Cohort 1; Placebo - Cohorts 2 and 3

SUMMARY:
This is a two-part, Phase 2, multi-center, randomized, double-blind, placebo-controlled, parallel design study of CA-008 (vocacapsaicin) vs. placebo injected/instilled during an elective TKA.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled, parallel design study evaluating, in a pilot stage of the study, up to 3 ascending dose level cohorts each evaluating a single dose of CA-008 vs. placebo injected/instilled during an elective TKA. Up to 54 subjects will be randomized in the pilot stage. During the optional second stage of the study, subjects will be randomized to one of either 2 or 3 CA-008 dose levels (to be determined) or placebo. The Sponsor made the decision not to proceed with the second stage.

ELIGIBILITY:
Key Inclusion Criteria:

1. Plan to undergo an elective primary unilateral total knee arthroplasty (TKA or knee replacement), without collateral procedure or additional surgeries.
2. Be a reasonably healthy adult aged 18 - 80 years old, inclusive, with a BMI ≤ 36 kg/m2 and American Society of Anesthesiology (ASA) physical Class 1, 2 or 3 at the time of randomization.
3. Males and females must abstain from intercourse, use acceptable birth control methods or be sterile or otherwise incapable of having children.
4. Be willing and able to sign the informed consent form (ICF)
5. Be willing and able to complete study procedures and pain scales and to communicate meaningfully in English. Be able and willing to return for outpatient follow up visits as required.

Key Exclusion Criteria:

1. In the opinion of the Investigator,

   1. have a concurrent painful condition, other than pain in the knee to be replaced, that may require pain treatment during the study period.
   2. have active skin disease or other clinically significant abnormality at the anticipated site of surgery that could interfere with the planned surgery.
2. Have a known allergy to chili peppers, capsaicin or the components of CA-008, ropivacaine, ketorolac, acetaminophen, fentanyl, hydromorphone, morphine or oxycodone.
3. Have significant medical, neuropsychiatric or other condition.
4. The following are considered disallowed medications:

   1. tolerant to opioids as defined
   2. capsaicin-containing products or foods.
   3. central nervous system active agent as an analgesic adjunct medication
   4. antiarrhythmics except beta-blockers, digoxin, warfarin, lithium, or aminoglycosides or other antibiotics for an infection
   5. parenteral or oral corticosteroids.
   6. antianginal, antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days or which is not expected to remain stable while participating in the study.
5. Have positive results on the alcohol breath/saliva test indicative of alcohol abuse or urine drug screen indicative of illicit drug use at screening, and/or prior to surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daneshvari Solanki, MD, Principal Investigator — First Surgical Hospital
Locations (1):
- HD Research, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One subject in Cohort 3, CA-008 15 mg had an adverse event before receiving treatment and was discontinued from the study without receiving study drug. This subject is not included in the results section
Groups:
- CA-008 5 mg (0.05 mg/mL) Cohort 1: Cohort 1 (5 mg), was prepared at 0.05 mg/mL CA-008
- Placebo - Cohort 1; Placebo - Cohorts 2 and 3: Placebo comparator identical in appearance to the investigational product, containing the same excipients as the active
- CA-008 10 mg (0.1 mg/mL) Cohort 2: Cohort 2 (10 mg), was prepared at 0.1 mg/mL CA-008
- CA-008 15 mg (0.15 mg/mL) Cohort 3: Cohort 3 (15 mg), was prepared at 0.15 mg/mL CA-008
Period: Overall Study
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo - Cohort 1 | CA-008 10 mg (0.1 mg/mL) Cohort 2 | CA-008 15 mg (0.15 mg/mL) Cohort 3 | Placebo - Cohorts 2 and 3
Started | 9 | 9 | 13 | 13 | 11
Completed | 9 | 9 | 12 | 11 | 10
Not Completed | 0 | 0 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The reason for the difference in the analysis population versus the number of participants in Participant Flow is due to the participant in CA-008 15 mg Cohort 3 who was randomized but not treated with study drug. This participant discontinued early from the study (on the same day of randomization) due to an adverse event.
Groups:
- Total: Total of all reporting groups
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo - Cohort 1 | CA-008 10 mg (0.1 mg/mL) Cohort 2 | CA-008 15 mg (0.15 mg/mL) Cohort 3 | Placebo - Cohorts 2 and 3 | Total
Number analyzed (Participants) | 9 | 9 | 13 | 12 | 11 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.62) | 61.4 (7.67) | 66.8 (7.30) | 67.0 (8.57) | 64.8 (7.26) | 65.2 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 8 | 6 | 4 | 29
  Male | 2 | 5 | 5 | 6 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 2 | 1 | 7
  Not Hispanic or Latino | 8 | 7 | 12 | 10 | 10 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 1 | 2 | 7
  White | 8 | 9 | 9 | 10 | 9 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 13 | 12 | 11 | 54

OUTCOME MEASURES:

1. Primary Outcome: Time-specific Mean Pain Intensity Scores (NRS) at Time 96 Hours for CA-008 vs. Placebo
Description: Primary Efficacy Endpoint for the Pilot Stage. Time-specific mean pain intensity scores at Time 96 hours for CA-008 vs. placebo based on a 10-point numerical rating scale (NRS) from 0-10 where 0 is no pain and 10 is the worst pain imaginable).
Time Frame: At 96 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo - Cohort 1 | CA-008 10 mg (0.1 mg/mL) Cohort 2 | CA-008 15 mg (0.15 mg/mL) Cohort 3 | Placebo - Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 13 | 12 | 11
scores on a scale | 3.8 (2.11) | 5.1 (2.85) | 4.9 (2.02) | 4.8 (3.47) | 5.5 (2.91)
Statistical Analysis 1: Comparison: CA-008 5 mg (0.05 mg/mL) Cohort 1 vs Placebo - Cohort 1; Test type: Superiority; p = 0.276, ANOVA
Statistical Analysis 2: Comparison: CA-008 10 mg (0.1 mg/mL) Cohort 2 vs Placebo - Cohorts 2 and 3; Test type: Superiority; p = 0.651, ANOVA
Statistical Analysis 3: Comparison: CA-008 15 mg (0.15 mg/mL) Cohort 3 vs Placebo - Cohorts 2 and 3; Test type: Superiority; p = 0.556, ANOVA

2. Primary Outcome: CA-008 Dose vs. Placebo Comparison: Area Under the Curve (AUC) 0 to 96 Hours
Description: Primary Efficacy Endpoint for Stage 2. Area Under the Curve (AUC) of the NRS current pain intensity scores from Time 0 hours to 96 hours at rest (AUC0 to 96h) where 0 is no pain and 10 is the worst pain imaginable for CA-008 compared to placebo. •
  During the inpatient stay, NRS at rest beginning with the PACU admission may be assessed once the subject is awake.
  The maximum is an NRS score of 10 x all 96 hours = 960 NRS units*hrs; the minimum is 0 x 96h = 0 NRS units*hrs
Time Frame: From 0 hours to 96 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: NRS units*hours
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo - Cohort 1 | CA-008 10 mg (0.1 mg/mL) Cohort 2 | CA-008 15 mg (0.15 mg/mL) Cohort 3 | Placebo - Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 13 | 12 | 11
NRS units*hours | 476.13 (182.315) | 593.93 (178.958) | 529.51 (147.247) | 532.14 (188.144) | 539.43 (217.047)
Statistical Analysis 1: Comparison: CA-008 5 mg (0.05 mg/mL) Cohort 1 vs Placebo - Cohort 1; Test type: Superiority; p = 0.136, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: CA-008 10 mg (0.1 mg/mL) Cohort 2 vs Placebo - Cohorts 2 and 3; Test type: Superiority; p = 0.649, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: CA-008 15 mg (0.15 mg/mL) Cohort 3 vs Placebo - Cohorts 2 and 3; Test type: Superiority; p = 0.608, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Subjects Who do Not Require Opioids
Description: Key Secondary Efficacy Endpoints for Stage 2. For each CA-008 dose vs. placebo comparison, percentage of subjects who do not require opioids.
Time Frame: Time 0 hours to Time 96 hours: Opioid Free 0 hours to 96 hours
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo - Cohort 1 | CA-008 10 mg (0.1 mg/mL) Cohort 2 | CA-008 15 mg (0.15 mg/mL) Cohort 3 | Placebo - Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 13 | 12 | 11
Participants | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: CA-008 5 mg (0.05 mg/mL) Cohort 1 vs Placebo - Cohort 1; Not estimable; Test type: Superiority; p = 0, Regression, Logistic — Not estimable; Not estimable; Odds Ratio (OR) = 0 — Not estimable
Statistical Analysis 2: Comparison: CA-008 10 mg (0.1 mg/mL) Cohort 2 vs Placebo - Cohorts 2 and 3; Not estimable; Test type: Superiority; p = 0, Regression, Logistic — Not estimable; Not estimable; Odds Ratio (OR) = 0 — Not estimable
Statistical Analysis 3: Comparison: CA-008 15 mg (0.15 mg/mL) Cohort 3 vs Placebo - Cohorts 2 and 3; Not estimable; Test type: Superiority; p = 0, Regression, Logistic — Not estimable; Odds Ratio (OR) = 0 — Not estimable

4. Secondary Outcome: Total Opioid Consumption (in Daily Oral Morphine Equivalents)
Description: Key Secondary Efficacy Endpoints for Stage 2. Mean total postoperative opioid consumption (in daily oral morphine equivalents) for CA-008 compared to placebo
Time Frame: OC from Time 0 hours to Time 96 hours: OC 0 hours to 96 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo - Cohort 1 | CA-008 10 mg (0.1 mg/mL) Cohort 2 | CA-008 15 mg (0.15 mg/mL) Cohort 3 | Placebo - Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 13 | 12 | 11
mg morphine equivalents | 244.17 (170.578) | 321.33 (137.462) | 242.77 (133.667) | 365.25 (201.161) | 280.36 (174.278)
Statistical Analysis 1: Comparison: CA-008 5 mg (0.05 mg/mL) Cohort 1 vs Placebo - Cohort 1; Test type: Superiority; p = 0.306, ANOVA
Statistical Analysis 2: Comparison: CA-008 10 mg (0.1 mg/mL) Cohort 2 vs Placebo - Cohorts 2 and 3; Test type: Superiority; p = 0.595, ANOVA
Statistical Analysis 3: Comparison: CA-008 15 mg (0.15 mg/mL) Cohort 3 vs Placebo - Cohorts 2 and 3; Test type: Superiority; p = 0.242, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 76 days for participants in the study. This was comprised of a screening period that could be up to 45 days and subsequent clinic visits through Day 29.
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information in this study did not differ from the clinicaltrials.gov definitions.
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo - Cohort 1 | CA-008 10 mg (0.1 mg/mL) Cohort 2 | CA-008 15 mg (0.15 mg/mL) Cohort 3 | Placebo - Cohorts 2 and 3
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/13 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 0/13 | 1/12 | 1/11
Other Adverse Events (participants affected / at risk) | 7/9 | 7/9 | 12/13 | 10/12 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 5 mg (0.05 mg/mL) Cohort 1 (N=9) | Placebo - Cohort 1 (N=9) | CA-008 10 mg (0.1 mg/mL) Cohort 2 (N=13) | CA-008 15 mg (0.15 mg/mL) Cohort 3 (N=12) | Placebo - Cohorts 2 and 3 (N=11)
Perforated ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CA-008 5 mg (0.05 mg/mL) Cohort 1 (N=9) | Placebo - Cohort 1 (N=9) | CA-008 10 mg (0.1 mg/mL) Cohort 2 (N=13) | CA-008 15 mg (0.15 mg/mL) Cohort 3 (N=12) | Placebo - Cohorts 2 and 3 (N=11)
Sinus tachycardia (Cardiac disorders) | 5 | 0 | 2 | 3 | 6
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 5 | 8 | 5 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4 | 5 | 2
Application site pain (General disorders) | 0 | 2 | 0 | 0 | 0
Instillation site induration (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 1
Perforated ulcer (General disorders) | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 2 | 4 | 2 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Incision site vesicles (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Allodynia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Post procedural drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 4 | 2
Hypotension (Vascular disorders) | 1 | 1 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT03731364/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT03731364/SAP_001.pdf